CLINICAL TRIAL: NCT02383290
Title: The Implementation of Pharmacogenomics Into Primary Care in British Columbia
Acronym: IPPC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: Genome British Columbia (Industry); Pfizer (Industry); Merck Sharp & Dohme LLC (Industry); Roche Pharma AG (Industry); GlaxoSmithKline (Industry); AstraZeneca (Industry); Health Research Foundation (Other); Janssen, LP (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: H14-02979
Record Dates: First submitted 2015-02-26; First posted 2015-03-09 (Estimated); Last update posted 2015-12-18 (Estimated); Status verified 2015-12

CONDITIONS: Pharmacogenetics

ARMS (1):
- Decision support (Experimental): This is a feasibility trial so all patients will give a saliva sample and the pharmacist/ Family Physician will use the decision support for generating prescription recommendations
  Interventions: Other: Decision support

INTERVENTIONS:
Other: Decision support — Saliva samples will be collected from each participant for genetic testing. A genetic report will be fed back to the research server, and into the Family Physicians/pharmacist's electronic record. The electronic record is linked to the UBC TreatGx computer; the next time the participant is seen by the Family Physician / Pharmacist personalized prescribing recommendations will be available for use.

SUMMARY:
Certain parts of the gene can predict how an individual person will respond to medication (pharmacogenetics). We will invite 250 individuals to give a sample of saliva. This sample will be sent to a laboratory for limited genomic analysis relating to pharmacogenetics. When personal data held by the participants, family physician, or pharmacist is joined with the genetic data personalized prescription recommendations are formed. The family physicians/pharmacists can view these recommendations through their electronic record. This should result in prescriptions that may be more beneficial and cause fewer adverse events.

DETAILED DESCRIPTION:
We wish to develop and test a decision support tool, TreatGx. Using genetic information (single nucleotide polymorphisms - SNPs) and patient biophysical characteristics this tool creates drug and dose recommendations.

Each year in Canada, there are approximately 200,000 severe adverse drug events, claiming 10,000 to 22,000 lives, and costing $13.7 to $17.7 billion. Physicians cannot predict whether a patient will gain the desired benefit from a prescribed medication or whether they will experience harmful side effects. Genetic tests may reduce this potential harm for many medications; however there is currently no way of incorporating genetic information into routine prescribing processes.

We see a need to pilot test a, genetic based, prescribing decision support (TreatGx) for feasibility and usability.

Five Family Physicians and one pharmacy will be invited to participate. They will be requested to identify a total of 250 adults with chronic diseases to participate in the study.

Each participant will be invited to give a saliva sample for the SNP test. This sample will be sent to the laboratory for genetic testing; whole genome testing is not being undertaken. We have identified from published evidence a small panel of SNPs that will give information to guide prescribing. A genetic report will be fed back into the family physician's or pharmacist's electronic health record. The electronic health record will be linked to TreatGx; the next time the participant is seen by the family physician/pharmacist prescribing recommendations will be available for use. The family physician will be able to use TreatGx to give the participant a prescription that is personalized.

We will track how many times the system is used, gain feedback on usability, record timing between receiving samples, time to the laboratory, time to analysis, and time to electronic record.

ELIGIBILITY:
Inclusion Criteria:

* People attending specified pharmacy or Family Physicians.
* Aged 18 years or over, with a chronic disease that requires medication.
* Chronic diseases include: gout, chronic obstructive pulmonary disease, depression, osteoarthritis, hypertension, hyperlipidemia, atrial fibrillation, asthma, osteoporosis and epilepsy.

Exclusion Criteria:

* Pregnant
* Breast feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2015-04; Primary Completion 2015-10 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Feasibility of recruitment (reported numbers of physicians and patients) | 6 months
Feasibility of obtaining SNP data (Number of lab reports generated) | 3 months
Feasibility of integrating SNP data into EMR (Number of lab reports integrated into EMR, time of sample to reach laboratory, time to analysis, and time to electronic record) | 3 months

SECONDARY OUTCOMES:
Use of decision support by family physicians and pharmacists (Number of times link is made to TreatGx by physicians/pharmacists) | 6 months
Reported usability of tool (User interviews) | 6 months
Estimated level of inappropriate prescribing (User interviews) | 6 months

REFERENCES:
- [Derived] Dawes M, Aloise MN, Ang JS, Cullis P, Dawes D, Fraser R, Liknaitzky G, Paterson A, Stanley P, Suarez-Gonzalez A, Katzov-Eckert H. Introducing pharmacogenetic testing with clinical decision support into primary care: a feasibility study. CMAJ Open. 2016 Sep 21;4(3):E528-E534. doi: 10.9778/cmajo.20150070. eCollection 2016 Jul-Sep. PMID 27730116